CLINICAL TRIAL: NCT03266991
Title: A Randomised Controlled Trial of a 12-dose Rifapentine and Isoniazid (RPT+INH) Regimen Using Direct Observed Therapy (DOT) Versus 6 Months of Daily Isoniazid for Latent Tuberculosis Infection (LTBI) in Socially Marginalised People
Brief Title: Treatment of Latent Tuberculosis in Socially Marginalised Citizens
Acronym: DOT-LTBI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Nina Breinholt Stærke, MD phd-student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A101A
Record Dates: First submitted 2017-08-11; First posted 2017-08-30 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2021-07

CONDITIONS: Compliance, Patient
MeSH Terms: conditions — Patient Compliance | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPT-INH (Experimental): Participants treated with weekly rifapentine and isoniazid for twelve weeks.
  Interventions: Drug: Rifapentine; Drug: Isoniazid
- control (Active Comparator): Participants treated with daily isoniazid for six months
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Rifapentine — Treatment with weekly rifapentine and isoniazid as Directly Observed Therapy in 12 weeks
  Other Names: isoniazid
  Arms: RPT-INH
Drug: Isoniazid — Treatment with daily isoniazid in 6 months

SUMMARY:
An open-label, randomised controlled trial comparing compliance to treatment for latent tuberculosis infection in socially marginalised citizens. Participants will be randomized to either daily isoniazid for 6 months or weekly rifapentine and isoniazid as directly observed therapy for twelve weeks.

DETAILED DESCRIPTION:
Eligible participants will be randomised to receive either daily isoniazid for 6 months with monthly visits for pill count, evaluation of adverse events and dispensing of isoniazid for the next month, or weekly doses of rifapentine and isoniazid for twelve weeks as direct observed therapy where the drugs are administered in the presence of a study nurse or doctor.

Control bloodsamples (ALAT, alkaline phosphatase, bilirubin, INR, haemoglobin, trombocytes and leukocyte differential count) will be taken at baseline and at least once during treatment in the rifapentine and isoniazid group and at least twice in the isoniazid-only group.

One year after treatment completion participants will be called in for evaluation for active tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Reporting to be homeless (independent of whether the person has an official address) or regularly seeking homeless shelters or public institutions to supply basic needs
* LTBI defined by positive IGRA test
* Found plausible by study doctor that the person has been exposed to tuberculosis within 2 years
* Aged 18 years or older

Exclusion Criteria:

* Previously treated for tuberculosis
* Pregnant or breastfeeding
* Active tuberculosis (evaluated by chest x-ray and examination by a trained doctor)
* Unable to give informed consent
* Tested positive for LTBI as part of contact investigation where the index case has or is suspected to have INH of RIF resistant TB
* Known HIV on antiretroviral treatment
* Porphyria
* Known allergy to rifamycins or isoniazid
* Known epilepsy
* Known liver disease causing affected liver parameters (ALAT, alkaline phosphatase, bilirubin, INR)
* Any lab abnormality, disease, concomitant medication or condition that, in the opinion of the investigator, excludes a person from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
adherence | 2 years
  adherence to treatment in the two groups measured by counting number of pills taken in each group.

SECONDARY OUTCOMES:
active tuberculosis | 5 years
  active tuberculosis within the study period. In case of suspected tuberculosis during the study the participant will be refered for examination by specialists. At 1 year follow-up participants will have a chest x-ray and physical examination by study doctor to screen for signs of active tuberculosis. If active tuberculosis is suspected further examinations will be performed by specialists.
adverse events | 2 years
  for both groups all adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wejse, MD PHD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Dept of Pulmonary Medicine, Aarhus
  - Dept of Pulmonary Medicine, Esbjerg

IPD SHARING:
Plan to Share IPD: No